CLINICAL TRIAL: NCT06089863
Title: Evaluation of the Effect of PAMPERO Rehabilitation Program in Collaboration With Patient Partner on the Symptom Intensity, Activity, and Quality of Life on Genetic and Degenerative Ataxia
Brief Title: Rehabilitation Program on Genetic and Degenerative Ataxia
Acronym: RAPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_0912
Record Dates: First submitted 2023-10-09; First posted 2023-10-18 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-10

CONDITIONS: Ataxia; Degenerative Disease; Genetic Disease
Keywords: Genetic ataxia; Degenerative ataxia; Rehabilitation; Cerebellar ataxia
MeSH Terms: conditions — Ataxia; Genetic Diseases, Inborn; Cerebellar Ataxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAMPERO program group (Experimental): This program is an intensive multidisciplinary program rehabilitation including Physical, Occupational, Speech, Psychomotor therapy and Adapted Physical Activity.
  Interventions: Other: PAMPERO program
- Usual Care intervention group (No Intervention): Usual Rehabilitation of the patient after the inclusion. 0 to 2 physical therapy sessions and 0 to 2 Speech therapy sessions each week usually constitute this program.
  This rehabilitation highly depends on the patients usual preferences. Some patients have no rehabilitation in the daily care while some have more.

INTERVENTIONS:
Other: PAMPERO program — This program is an intensive multidisciplinary program rehabilitation including Physical, Occupational, Speech, Psychomotor therapy and Adapted Physical Activity. The duration of this program is 5 weeks and each week is divided as follow :
  * 5 hours of physical therapy : individual session with the objective to improve the dynamic balance and coordination on the aim to gain confidence of moving, gripping capacity and interaction with object
  * 5 hours of Adapted Physical activity : group session to promote pairing with muscle building priority
  * 1 hour of Speech therapy : group session to educate and promote prevention strategy about dysphagia rick
  * 2 hours of Occupational therapy : group session to bring adaptive solution of autonomy lost with material propose, home organisation or gesture
  * 2 hours of Hydrotherapy : group session activity performed in water to assist rehabilitation
  Arms: PAMPERO program group

SUMMARY:
Cerebellar ataxia is a pathology linked to the lesion of the cerebellum or the afferent and/or efferent cerebellar pathways. The aetiology can be an acquired cerebral lesion, following a chemical poisoning or a genetic degenerative lesion (for example : Friedreich's ataxia, spinocerebellar ataxias, etc.). As reported by the latest estimate available, genetic degenerative cerebellar ataxias affect approximately 6,000 patients in France (Orpha.net). Symptoms suffered by ataxic patients are : problems and gait disorders along with difficulties in coordination resulting in ataxia, uncoordinated movements.

These symptoms cause a decrease in the quality of life on patients with spinocerebellar ataxia. The symptoms improvement linked to the cerebellar syndrome is based on rehabilitation that can be supplemented by use of technical aids. Current scientific knowledge confirms that intensive rehabilitation by physiotherapy and occupational therapy in patients with degenerative ataxias improves cerebellar symptoms. Nevertheless, the choice rehabilitation technique stay at the appreciation of the therapist.

From the observation, the investigators have designed an intensive multidisciplinary rehabilitation program, called PAMPERO, with partner patients member of two genetic degenerative ataxia patient organisations. This 5-weeks program has been used in clinic during 3 years on 28 patients. It appears to be the only one in France.

The preliminary results show a positive effect on ataxia symptom. Nevertheless, the duration of the benefice over time and the effect on the quality of life stay unknown.

However, the quality of life is mainly affected by the participation restriction due to the risk of falling. The most frequent complaint from partner patient is the diminution of the social interaction resulting of the incapacity to move without risk.

The present protocol aimed at evaluating the Rehabilitation Program in collaboration with partner patient on the symptom intensity, activity and quality of life on genetic and degenerative ataxia.

This PAMPERO program's effect will be assessed by comparing the difference of Intensity of symptom measured by to Scale for the Assessment and Rating of Ataxia (SARA) at inclusion and 3 months after the end of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Patients with genetic and degenerative cerebellar ataxia
* Diagnostic of cerebellar ataxia confirmed by anatomic MRI
* Affiliated to a social insurgence regime or similar
* Patients who have given their free, informed and express consent
* Walking patients (who can walk unsupervised on flat ground with the help of proper technique : categories greater than 4 on the New Functional Ambulation Classification scale)

Non inclusion Criteria:

* Patients who have already benefited from a hospitalization of more than 3 weeks for rehabilitation during the last 12 months
* Patients participating simultaneously in another research whose objective would be the evaluation of a therapy, medicinal or not, likely to improve neurological or functional recovery
* Pregnants, parturient or breastfeeding
* Patients deprived of their liberty by a judicial or administrative decision
* Psychiatric care patients
* Patients admitted to Patients admitted to a health or social establishment for purposes other than research for purposes other than research
* Major patients protected by the Law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | Inclusion ; 3 months after the end of rehabilitation
  Intensity of symptom measured by to Scale for the Assessment and Rating of Ataxia (SARA). Scores are from 0 to 42. An higher score is associated with a worse outcome.

SECONDARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia (SARA) | Inclusion ; Immediately or 1 week after the end of rehabilitation ; 6 months after the end of rehabilitation
  Intensity of symptom measured by to Scale for the Assessment and Rating of Ataxia (SARA). Scores are from 0 to 42. An higher score is associated with a worse outcome.
Score of the Mini-BESTest scale | Inclusion ; Immediately or 1 week after the end of rehabilitation ; 3 months after the end of rehabilitation ; 6 months after the end of rehabilitation
  Measure of the balance evaluate by Mini-BESTest scale (Mini-Balance Evaluation Systems Test). Scores are from 0 to 28. An higher score is associated with a better outcome.
Eyes open postural surface | 5 weeks
  Measure of the balance evaluate by the Eyes open postural surface
Displacement length of the center of mass as a function of time eyes open | 5 weeks
  Measure of the balance evaluated by the displacement length of the center of mass as a function of time eyes open
Scale of Short Falls Efficacy Scale International (Short FES-I) | Inclusion ; Immediately or 1 week after the end of rehabilitation ; 3 months after the end of rehabilitation ; 6 months after the end of rehabilitation
  Fear of fall evaluated by to Scale of Short Falls Efficacy Scale International (Short FES-I). Scores are from 7 to 28. An higher score is associated with a worse outcome.
Number of weekly steps | Inclusion ; Immediately or 1 week after the end of rehabilitation ; 3 months after the end of rehabilitation ; 6 months after the end of rehabilitation
  Number of steps during one week continuously measured by actimeter ActiGraph wGT3X-BT with EUROCOC (European Certificate of Conformity)
Time of weekly sedentary activity | Inclusion ; Immediately or 1 week after the end of rehabilitation ; 3 months after the end of rehabilitation ; 6 months after the end of rehabilitation
  Time in minutes/day of sedentary activity during one week continuously measured by actimeter ActiGraph wGT3X-BT with EUROCOC
Light, moderate and vigorous weekly activity | Inclusion ; Immediately or 1 week after the end of rehabilitation ; 3 months after the end of rehabilitation ; 6 months after the end of rehabilitation
  Light, moderate and vigorous activity during one week continuously measured by actimeter ActiGraph wGT3X-BT with EUROCOC
Short Form Health Survey (SF-36) | Inclusion ; Immediately or 1 week after the end of rehabilitation ; 3 months after the end of rehabilitation ; 6 months after the end of rehabilitation
  Measure of the quality of life evaluate by Short Form Health Survey (SF-36). Scores are from 0 to 100. An higher score is associated with a better outcome.
Number of falls during the study | 4 weeks ; up to 3 months ; up to 6 months
  Risk of falling evaluated by the number of falls during and outside the rehabilitation normalized on 4 weeks
Number of patients who completed the entire PAMPERO program | 5 weeks
  Number of patients who completed the entire PAMPERO program (5 weeks)
Number of patients who stopped PAMPERO program | 5 weeks
  Number of patients who stopped PAMPERO program
Time to occurrence of PAMPERO program stops | 5 weeks
  Time to occurrence of PAMPERO program stops
Reasons of PAMPERO program stops | 5 weeks
  Reasons of PAMPERO program stops

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de Rééducation Fonctionnelle (S.S.R.) Val Rosay, Saint-Didier-au-Mont-d'Or
  - Service de Médecine Physique et Réadaptation (M.P.R) de l'Hôpital Bellevue, Saint-Etienne
  - Service de Rééducation Fonctionnelle (S.S.R.) de l'Hôpital Henry Gabrielle Hospices Civils de Lyon, Saint-Genis-Laval